CLINICAL TRIAL: NCT05666492
Title: "Platelet Rich Plasma for the Management of Post-Viral Olfactory Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thomas Jefferson University (Other)
Collaborators: Monell Chemical Senses Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22D.470
Record Dates: First submitted 2022-08-15; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Olfactory Disorder; Olfaction Disorders
Keywords: Olfaction; Smell
MeSH Terms: conditions — Olfaction Disorders; Anosmia | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled randomized control trial
Who Masked: Participant
Masking Description: Subjects will be randomized into test or control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Less than 12 months PRP- Test (Experimental): Patients randomized into the less than 12 months PRP arm will receive 3 doses of topical PRP each month apart and their sense of smell will be assessed during each visit followed by a monthly remote assessment of smell from home.
  Interventions: Other: Platelet rich plasma
- Less than 12 months placebo- control (Placebo Comparator): Patients randomized into the less than 12 months placebo arm will receive saline topically every month apart and their sense of smell will be assessed during each visit followed by a monthly remote assessment of smell from home.
  Interventions: Other: Saline
- More than 12 months PRP- Test (Experimental): Patients randomized into more than 12 months PRP arm will receive 3 doses of topical PRP each month apart and their sense of smell will be assessed during each visit followed by a monthly remote assessment of smell from home.
  Interventions: Other: Platelet rich plasma
- More than 12 months Placebo- Control (Placebo Comparator): Patients randomized into the less than 12 months placebo arm will receive saline topically every month apart and their sense of smell will be assessed during each visit followed by a monthly remote assessment of smell from home.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Platelet rich plasma — Platelet-rich plasma will be placed on the olfactory epithelium topically.
  Arms: Less than 12 months PRP- Test; More than 12 months PRP- Test
Other: Saline — Saline will be placed on the olfactory epithelium topically.
  Arms: Less than 12 months placebo- control; More than 12 months Placebo- Control

SUMMARY:
SARS COV-19 has resulted in prolonged olfactory dysfunction in many patients. The investigators aim to compare the effect of topical platelet-rich plasma (test) vs saline (placebo) in patients with covid-related post-viral olfactory dysfunction.

DETAILED DESCRIPTION:
The investigators hypothesize that the use of topical PRP will improve smell identification, threshold, and smell-related quality of life in comparison to a placebo.

This study will provide critical information for a promising new treatment of olfactory dysfunction with the highest level of evidence, in a randomized, placebo-controlled trial. Preliminary results from an ongoing pilot study investigating topical PRP is the basis for the hypothesis.

By investigating the efficacy of topical PRP in smell restoration, the investigators will provide a less-invasive way to deliver this autologous product. A randomized trial will set a precedent for the use of this treatment to serve a growing population of patients affected with post-COVID olfactory dysfunction. Over a period of one year, participants with post-viral olfactory dysfunction will be randomly assigned to a test or control group and will visit the clinic monthly for three months to receive PRP or saline based on their randomized group. This will be followed by 9 months of at-home electronic visits. At each visit both the test and control groups will undergo smell testing and will fill quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suffering from either post-viral or post-COVID smell loss of any duration, without a history of nasal surgery, nasal polyposis, chronic rhinosinusitis, or intranasal tumors
* Patients who are post-COVID must report at least a positive home test on history
* Patients with post-viral etiology must have recall of a viral illness that immediately preceded smell loss

Exclusion Criteria:

* History of olfactory dysfunction predating COVID-19 infection
* History of trauma, previous surgery, or obstructive cause of OD (nasal polyps, chronic rhinosinusitis)
* Pregnancy
* Patients who are unable to provide consent
* Patients with known bleeding disorders
* Patients with known malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
Effect of PRP on smell identification | Every month for 12 months
  Investigate the effect of topical PRP on olfaction via smell identification testing using a brief smell identification test (B-SIT). The change in smell identification with PRP or placebo over time will be assessed using B-SIT, a validated 12-odorant scratch-and-sniff questionnaire. The maximum possible score is 12, and the minimum score is 0. A score greater than or equal to 8 is considered normal olfaction, while a score lesser than three should raise a suspicion of malingering. Hence a higher score implies better outcomes.
Effect of PRP on smell intensity | Every month for 12 months
  Investigate the effect of topical PRP on olfaction via smell identification testing using SCENTinel smell test.
  The SCENTinel test assesses for odor identification and the threshold of identification. Every month the participant is provided with one SCENTinel card - a QR-coded Lift'n'smell card containing a single target odorant and two blank odorants. The QR code leads to an electronic questionnaire the subject must fill out. Results with less than 40% Odor threshold are considered olfactory dysfunction. Hence a higher score implies better outcomes. The change in participants' threshold of identification will be assessed monthly over a year.
Effect of PRP on smell related quality of life | Every month for 12 months
  Investigate and compare the effect of topical PRP vs saline on quality of life participants using the Questionnaire of olfactory disorders negative statements only (QODNS) scale.
  QODNS scale has 17 questions with each question scored between 0 to 3. The maximum score is 51 and the minimum score is 0 with higher scores being inversely related to the quality of life ie a higher score implies worse quality of life. The change in quality of life will be assessed monthly over one year.

SECONDARY OUTCOMES:
Natural course of covid related olfactory dysfunction | 12 months from clinic visit
  Investigate the natural course of post-COVID / post-viral olfactory dysfunction in patients treated with placebo for the study by comparing the smell test.

CONTACTS AND LOCATIONS:
Overall Officials: David Rosen, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan CH, Mundy DC, Patel ZM. The use of platelet-rich plasma in treatment of olfactory dysfunction: A pilot study. Laryngoscope Investig Otolaryngol. 2020 Feb 21;5(2):187-193. doi: 10.1002/lio2.357. eCollection 2020 Apr. PMID 32337347
- [Background] Yasak AG, Yigit O, Araz Server E, Durna Dastan S, Gul M. The effectiveness of platelet-rich plasma in an anosmia-induced mice model. Laryngoscope. 2018 May;128(5):E157-E162. doi: 10.1002/lary.27029. Epub 2017 Dec 15. PMID 29243256
- [Background] Mattos JL, Edwards C, Schlosser RJ, Hyer M, Mace JC, Smith TL, Soler ZM. A brief version of the questionnaire of olfactory disorders in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Oct;9(10):1144-1150. doi: 10.1002/alr.22392. Epub 2019 Aug 20. PMID 31430061
- [Background] Mavrogeni P, Kanakopoulos A, Maihoub S, Krasznai M, Szirmai A. Anosmia treatment by platelet rich plasma injection. Int Tinnitus J. 2017 Apr 19;20(2):102-105. doi: 10.5935/0946-5448.20160019. PMID 28452719